CLINICAL TRIAL: NCT00706095
Title: An Open-label, Parallel Group Study to Explore the Pharmacokinetics of Eribulin Mesylate (E7389) in Patients With Advanced Solid Tumors and Normal or Reduced Hepatic Function According to the Child-Pugh System
Brief Title: Study Of Eribulin (E7389) In Patients With Advanced Solid Tumors And Normal Or Reduced Hepatic Function As Per Child-Pugh System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-E044-108
Record Dates: First submitted 2008-02-04; First posted 2008-06-27 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Cancer
Keywords: Cancer; advanced solid tumors
MeSH Terms: conditions — Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- E7389 1.4 mg/m^2 (Experimental)
  Interventions: Drug: E7389
- E7389 1.1 mg/m^2 (Experimental)
  Interventions: Drug: E7389
- E7839 0.7 mg/m^2 (Experimental)
  Interventions: Drug: E7389

INTERVENTIONS:
Drug: E7389 — E7389 Intravenous injection starting dose on Day 1 is 1.4 mg/m^2 for normal hepatic function.
  Other Names: Eribulin mesylate
  Arms: E7389 1.4 mg/m^2
Drug: E7389 — E7389 Intravenous injection starting dose on Day 1 is 1.1 mg/m^2 for mild hepatic impairment (Child-Pugh A)
  Other Names: Eribulin mesylate
  Arms: E7389 1.1 mg/m^2
Drug: E7389 — E7389 Intravenous injection starting dose on Day 1 is 0.7 mg/m^2 for moderate hepatic impairment (Child-Pugh B)
  Other Names: Eribulin mesylate
  Arms: E7839 0.7 mg/m^2

SUMMARY:
This is an open-label, three-parallel group pharmacokinetic study. Patients with advanced solid tumors will be assigned to one of three groups to receive I.V. doses of eribulin (E7389). The three groups are: normal hepatic function, mild hepatic impairment (Child-Pugh A) and moderate hepatic impairment (Child-Pugh B) according to the Child-Pugh System for classifying hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically or cytologically confirmed advanced solid tumor that has progressed following standard therapy or for which no standard therapy exists (including surgery or radiation therapy)
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
4. Life expectancy of ≥ 3 months
5. Adequate renal function as evidenced by serum creatinine ≤ 2.0 mg/dL or calculated creatinine clearance ≥ 40 mL/minute (min) per the Cockcroft and Gault formula.
6. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, hemoglobin ≥ 10.0 g/dL (a hemoglobin <10.0 g/dL is acceptable if it is corrected by growth factor or transfusion), and platelet count ≥ 100 x 10^9/L
7. Patients willing and able to comply with the study protocol for the duration of the study
8. Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Additional Inclusion Criteria for the Group of Patients with No Hepatic Impairment:

* All the general inclusion criteria listed above plus: Normal hepatic function as evidenced by bilirubin ≤ 34 μmol/l (≤2.0 mg/dL) and alkaline phosphatase, alanine transaminase (ALT), and aspartate transaminase (AST) ≤3 times the upper limits of normal (ULN) (in the case of liver metastases ≤5 x ULN), or in the case of bone metastases, the liver specific alkaline phosphatase ≤3 times the upper limits of normal (ULN), and in the case of concomitant liver metastases, ≤5 x ULN.

Additional Inclusion Criteria for the Group of Patients with Hepatic Impairment:

* All the general inclusion criteria listed above plus:

  * Mild (Child-Pugh A) or moderate (Child-Pugh B) hepatic dysfunction according to the Child-Pugh scoring system criteria, where patients with laboratory values within normal ranges will not be included in the Child-Pugh A category
  * Or, Moderate hepatic dysfunction (Child-Pugh B) according to the Child-Pugh scoring system criteria

Exclusion Criteria:

1. Patients who have received any of the following treatments within the specified period before E7389 treatment start:

   1. Chemotherapy, radiation, biological therapy within 3 weeks.
   2. Hormonal therapy within 1 week.
   3. Any investigational drug within 4 weeks.
2. Patients with any clinically significant laboratory abnormality except for those parameters influenced by hepatic impairment.
3. Patients with severe (Child-Pugh C) hepatic dysfunction according to the Child-Pugh scoring system.
4. Patients with encephalopathy ≥ Grade 1.
5. Patients receiving any drug known to induce or inhibit CYP3A4 activity. Clinically significant drugs are listed in a comprehensive list that can be found at http://medicine/iupui.edu/flockhart/table.htm.
6. Patients, who require therapeutic anti-coagulant therapy other than for line patency with warfarin or related compounds and cannot be changed to heparin-based therapy, are not eligible.
7. Women who are pregnant or breast-feeding; women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test; women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator. Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
8. Fertile men who are not willing to use contraception or fertile men with a female partner who are not willing to use contraception
9. Severe/uncontrolled intercurrent illness/infection.
10. Significant cardiovascular impairment (history of congestive heart failure > New York Heart Association [NYHA] Grade II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia).
11. Patients with organ allografts requiring immunosuppression (not including blood and blood components transfusions).
12. Patients with known positive HIV status.
13. Patients with brain or subdural metastases are not eligible, unless they are stable and have completed local therapy and have discontinued the use of corticosteroids for this indication for at least four weeks before starting treatment with E7389.
14. Patients with meningeal carcinomatosis.
15. Patients with a hypersensitivity to halichondrin B and/or halichondrin B-like compounds.
16. Patients who participated in a prior E7389 clinical trial.
17. Patients with preexisting neuropathy > Grade 2.
18. Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. JHM Schellens, Principal Investigator — National Cancer Institute-Antoni van Leuwenhoek Hospital
Locations (2):
- Netherlands (2):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Utrecht Medical Centre, Utrecht

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 2 centers in The Netherlands during the period of Feb 2008 to Jan 2010.
Groups:
- E7389 1.4 mg/m^2: E7389 Intravenous injection starting dose on Day 1 is 1.4 mg/m^2 for normal hepatic function.
- E7389 1.1 mg/m^2: E7389 Intravenous injection starting dose on Day 1 is 1.1 mg/m^2 for mild hepatic impairment (Child-Pugh A)
- E7389 0.7 mg/m^2: E7389 Intravenous injection starting dose on Day 1 is 0.7 mg/m^2 for moderate hepatic impairment (Child-Pugh B)
Period: Overall Study
Arm/Group | E7389 1.4 mg/m^2 | E7389 1.1 mg/m^2 | E7389 0.7 mg/m^2
Started | 6 | 7 | 5
Completed | 0 | 0 | 0
Not Completed | 6 | 7 | 5
Not completed — Progressive Disease | 4 | 5 | 3
Not completed — Clinical Progression | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E7389 1.4 mg/m^2 | E7389 1.1 mg/m^2 | E7389 0.7 mg/m^2 | Total
Number analyzed (Participants) | 6 | 7 | 5 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 60.2 (5.98) | 59.9 (4.88) | 65.2 (2.68) | 61.4 (5.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 7
  Male | 5 | 2 | 4 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White | 6 | 7 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean (SD) Pharmacokinetic (PK) Parameter Area Under Concentration Time Curve From Zero to Infinity (AUC0-oo)
Time Frame: Pre-dose (-0.5h); post-dose at 15 min, 30 min, 60 min, 2 hrs, 4 hrs, 6 hrs, 10 hrs, 24 hrs, 48 hrs, 72hrs, 96 hrs, 120 hrs and 144 hours.
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | E7389 1.4 mg/m^2 | E7389 1.1 mg/m^2 | E7389 0.7 mg/m^2
Number analyzed (Participants) | 6 | 7 | 5
ng*hr/mL | 600 (267.1) | 731 (288.3) | 720 (407.4)

2. Primary Outcome: Mean (SD) Pharmacokinetic (PK) Parameter Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | E7389 1.4 mg/m^2 | E7389 1.1 mg/m^2 | E7389 0.7 mg/m^2
Number analyzed (Participants) | 6 | 7 | 5
ng/mL | 186 (67.4) | 147 (47.6) | 113 (47.2)

3. Primary Outcome: Best Overall Response Per Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Defined as the best response from the start of treatment until disease progression or recurrence. Lesions measured by computed tomography (CT) scan and magnetic resonance imaging (MRI). Objective response rate: complete response (CR-disappearance of all lesions)+ partial response (PR-30% decrease in lesion diameter), Progressive Disease (PD-20% increase in lesion diameter), stable disease (SD-neither shrinkage nor increase of lesions).
Time Frame: throughout the study and up to 30 days after the last dose of study drug
Population: ITT Population
Measure: Number; unit: Number of Participants
Arm/Group | E7389 1.4 mg/m^2 | E7389 1.1 mg/m^2 | E7389 0.7 mg/m^2
Number analyzed (Participants) | 6 | 7 | 5
Number of Participants
  Best Overall Response - Complete Response | 0 | 0 | 0
  Best Overall Response - Partial Response | 0 | 0 | 0
  Best Overall Response - Stable Disease | 4 | 1 | 4
  Best Overall Response - Progressive Disease | 2 | 5 | 1
  Best Overall Response - Missing | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | E7389 1.4 mg/m^2 | E7389 1.1 mg/m^2 | E7389 0.7 mg/m^2
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/7 | 3/5
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 1.4 mg/m^2 (N=6) | E7389 1.1 mg/m^2 (N=7) | E7389 0.7 mg/m^2 (N=5)
Duodenal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Esophageal Varices Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 1.4 mg/m^2 (N=6) | E7389 1.1 mg/m^2 (N=7) | E7389 0.7 mg/m^2 (N=5)
Nausea (Gastrointestinal disorders) | 3 | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 4 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal Distention (Gastrointestinal disorders) | 0 | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 1 | 1
Melena (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 2 | 6 | 3
Edema Peripheral (General disorders) | 0 | 1 | 2
Pyrexia (General disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscular Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Weight Decreased (Investigations) | 1 | 2 | 2
Blood Bilirubin Increased (Investigations) | 0 | 2 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 1
Blood Creatinine Increased (Investigations) | 0 | 2 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 4
Dysgeusia (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Confusional State (Psychiatric disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No